CLINICAL TRIAL: NCT03959839
Title: Endoscopic Submucosal Dissection Versus Local Laparoscopic Surgical Resection (Transanal Minimally Invasive Surgery [TAMIS] / Transanal Endoscopic Operation [TEO]) In Early Rectal Neoplasias. Multicentric and Randomized Clinical Trial
Brief Title: Endoscopic Submucosal Dissection vs Local Laparoscopic Surgical Resection (TAMIS/TEO) in Early Rectal Neoplasias
Acronym: DSETAMIS2018
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Alberto Herreros de Tejada Echanojáuregui (Other)
Collaborators: Spanish Society of Digestive Endoscopy (Other)
Responsible Party: Sponsor-Investigator, Dr. Alberto Herreros de Tejada Echanojáuregui, Principal Investigator, Puerta de Hierro University Hospital
Organization: Puerta de Hierro University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSETAMIS-2018
Record Dates: First submitted 2019-05-16; First posted 2019-05-22 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Rectal Neoplasms
Keywords: Early Rectal Neoplasms; ESD; TAMIS; TEO; Recurrence; R0; Safety
MeSH Terms: conditions — Rectal Neoplasms; Recurrence | interventions — Transanal Endoscopic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endoscopic Treatment (Experimental): Rectal Endoscopic Submucosal Dissection
  Interventions: Procedure: ESD
- Minimally Invasive Laparoscopic Local Surgical Treatment (Experimental): Transanal Minimally Invasive Surgery (TAMIS) or Transanal Endoscopic Operation (TEO)
  Interventions: Procedure: TAMIS; Procedure: TEO

INTERVENTIONS:
Procedure: ESD — Rectal Endoscopic Submucosal Dissection
  Arms: Endoscopic Treatment
Procedure: TAMIS — Transanal Minimally Invasive Surgery
  Arms: Minimally Invasive Laparoscopic Local Surgical Treatment
Procedure: TEO — Transanal Endoscopic Operation
  Arms: Minimally Invasive Laparoscopic Local Surgical Treatment

SUMMARY:
A multicenter non-inferiority randomized clinical trial to compare Endoscopic treatment (ESD) and Minimally Invasive Laparoscopic Local Surgical Treatment (TAMIS or TEO) for early rectal neoplastic lesions (adenoma & T1CRC) Primary aim: To compare the long-term local recurrence rate (12 months after the procedure)

Secondary aims:

Compare en-bloq resection rate, R0 resection, time per procedure, short-term recurrence rate, safety (rate of complications), morbidity and cost-effectiveness analyses.

DETAILED DESCRIPTION:
A multicenter non-inferiority randomized clinical trial is proposed to compare two types of treatment for early rectal neoplastic lesions. Study arms:

1. Endoscopic treatment: Endoscopic Submucosal Dissection (ESD)
2. Minimally invasive laparoscopic local surgical treatment: Transanal Minimally Invasive Surgery (TAMIS) or Transanal Endoscopic Operation (TEO).

Aims:

Primary aim: To compare the long-term local recurrence rate (12 months after the procedure) of rectal lesions after ESD vs Surgical treatment (TAMIS/TEO).

Secondary aims: Both arms of the study are compared according to other efficacy-related variables (en-bloq resection rate, R0 resection, time per procedure, short-term recurrence rate [6 months]), safety (rate of complications), morbidity (comparing different specific indexes: Wexner index, EQ-5L-5D, etc) and cost-effectiveness analyses (QALY).

Inclusion criteria:

* Patients older than 18 y/o
* Non-pedunculated rectal lesions (sessile 0-Is or flat 0-II) greater than 20 mm in diameter.
* The edges of the lesion should be more than 3 cm from the external anal margin and up to 14 cm from it.
* Circumferential involvement <50%

Exclusion criteria:

* Patients who refuse to participate.
* Diagnosis of inflammatory bowel disease with rectal involvement.
* Pregnant.
* Anorectal fibrosis due to previous anorectal surgery.
* Lateral Spreading Lesions (LST classification) Granular Homogeneous type
* Lesions greater than 50 mm when there is suspicion of advanced histology (Kudo Vi superficial pattern).
* Rectal lesions of any size with high suspicion of deep submucosal invasion or locoregional lymph node involvement, either in the diagnostic colonoscopy (Kudo Vn crypt pattern, NICE 3 pattern, Sano IIIB pattern) or by complementary imaging tests (rectal EUS/Pelvic MRI)
* Existence of synchronous colorectal lesions that require other surgical treatment in any case.

N-size estimation:

Assuming a global rate of long-term local recurrence in rectal lesions treated by TAMIS/TEO or ESD of 2.5% (using the data available in the medical literature), considering a non-inferiority limit of 10%, power of 80% (Beta error 0.2, alpha error 0.05) and assuming a loss of patients during the follow-up around 10%, 34 patients per group are required.

Follow-up and Information collect:

The follow-up will be of 1 year from the date of the intervention and the visits in which the information to be analyzed will be collected are adjusted to the usual clinical practice.

The data would be registered using the on-line database system for medical research RedCap.

Other information:

The entire protocol of this study has been approved by de Ethical Committee on Clinical Research of the Puerta de Hierro University Hospital.

The study counts with a Civil Responsibility Insurance policy.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 y/o
* Non-pedunculated rectal lesions (sessile 0-Is or flat 0-II) greater than 20 mm in diameter.
* The edges of the lesion should be more than 3 cm from the external anal margin and up to 14 cm from it.
* Circumferential involvement <50%

Exclusion Criteria:

* Patients who refuse to participate.
* Diagnosis of inflammatory bowel disease with rectal involvement.
* Pregnant.
* Anorectal fibrosis due to previous anorectal surgery.
* Lateral Spreading Lesions (LST classification) Granular Homogeneous type
* Lesions greater than 50 mm when there is suspicion of advanced histology (Kudo Vi superficial pattern).
* Rectal lesions of any size with high suspicion of deep submucosal invasion or locoregional lymph node involvement, either in the diagnostic colonoscopy (Kudo Vn pit pattern, NICE 3 pattern, Sano IIIB pattern) or by complementary imaging tests (rectal EUS/Pelvic MRI)
* Existence of synchronous colorectal lesions that require other surgical treatment in any case.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
local recurrence rate | 12 months
  presence of remaining neoplastic tissue in resection site

SECONDARY OUTCOMES:
En-bloq resection rate | 1 hour
  Single piece of resection specimen
R0 resection rate | 1 hour
  Free margin of neoplastic tissue both laterally and deep
Time per procedure | 1 hour
  The length of the procedure expressed in minutes
Length of hospital stay | 1 hour
  Days of hospital stay
Early complications rate | 1 hour
  Registration of any deviations on the normal postoperative period in the first 24 hours
Delayed complications rate | 1 hour
  Registration of any deviations on the normal postoperative period after the first 24 hours and up to 30 days after the procedure
Morbidity | 12 months
  Changes in patients' quality of life using validated scores (both, specific and non-specific)
Cost-effectiveness analyses (QALY) | 12 months
  Cost-effectiveness analyses usin QALYs
Short-term local recurrence rate | 6 months
  Presence of remaining neoplastic tissue in resection site

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Albéniz, MD, PhD, Study Director — Complejo Hospitalario de Navarra
Locations (3):
- Spain (3):
  - Hospital de Sant Joan Despí Moisès Broggi, Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Frutos Rosa D, Alonso Sebastian I, Barquero Declara D, Badia Closa J, Nogales O, Jimenez Gomez LM, Santiago Garcia J, Valentin Gomez F, Royuela Vicente A, Sanchez Movilla A, Albeniz E, Herreros de Tejada Echanojauregui A; Mucosal Resection; Third-Space Endoscopy Working Group from the Spanish Society of Gastrointestinal Endoscopy. A Randomized Trial of Endoscopic Submucosal Dissection vs Transanal Minimally Invasive Surgery in Early Rectal Neoplasms: DSETAMIS-2018 Study. Gastroenterology. 2026 Jan;170(1):161-173. doi: 10.1053/j.gastro.2025.07.029. Epub 2025 Jul 30. PMID 40749854